CLINICAL TRIAL: NCT03799406
Title: Does Oral Vitamin D Supplementation in Egyptian Infants With Acute Bronchiolitis Improve the Outcome? A Double Blind Randomized Controlled Trial
Brief Title: Vitamin D Supplementation for Acute Bronchiolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amal Osman, Lecturer of Pediatrics, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS/16.01.38
Record Dates: First submitted 2018-12-29; First posted 2019-01-10 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Bronchiolitis
Keywords: Acute bronchiolitis; Vitamin D; Modified Tal score; Randomized; Controlled trial
MeSH Terms: conditions — Bronchiolitis | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): cholecalciferol at dose of 100 IU/Kg/day
  Interventions: Drug: Cholecalciferol
- Placebo group (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Therapeutic trial of vitamin D supplementation during acute episode of bronchiolitis
  Other Names: Vitamin D
  Arms: Intervention group
Other: Placebo — Placebo supplementation during acute episode of bronchiolitis
  Arms: Placebo group

SUMMARY:
This study was conducted to evaluate the effect of oral vitamin D supplementation on the clinical course of acute bronchiolitis, and to investigate whether vitamin D deficiency among infants who required hospital-based care for bronchiolitis is associated with the severity of the acute episode.

DETAILED DESCRIPTION:
This is a double blind randomized controlled trial which was conducted on 60 infants who required hospital-based care for acute bronchiolitis. The patients were recruited in the period from October 2018 to January 2019. Informed consents were obtained from all caregivers, and approved by Institutional Research Board of our University.

The diagnosis of acute bronchiolitis was based on a first episode of respiratory distress with wheezing and/ or crackles, preceded by an infection of the upper airways (rhinorrhea, coryza, cough, fever). Disease severity was evaluated using Modified-Tal scoring systems for bronchiolitis, since it is repeatable and can reliably be used in research and clinical practice

Sample size:

Our hospital data have shown that the mean LOS for cases admitted with acute bronchiolitis was 3 ± 2 days. Assuming a reduction in length of hospital stay by 50% and study power of 80% to detect a clinical significance (α error) of 0.05 between interventional groups, we calculated a sample size of 30 patients in each treatment group.

Randomization and Enrollment:

Patients were randomized to receive vitamin D3 treatment [100 IU/Kg/day in acute bronchiolitis] (vitamin D group) or placebo (placebo group) all through the period of admission as a previous cohort observational study has postulated that vitamin D daily dose close to 100 IU/kg body weight is favorable for infants up to age 12 months. Both groups were equal in number. Both vitamin D3 and placebo were in drop form and were identical in shape and nearly the same taste and color. The assignments were kept in sealed envelopes till data analysis. The randomization and allocation process were done by a higher nursing staff blinded to the study. Throughout the study, the medical staff, and parents were blind to assignments.

All patients were hospitalized and received treatment. The treatment consisted of intravenous fluids, oxygenation, and antipyretics if needed, and nebulized hypertonic saline. Nebulized adrenaline or salbutamol was added in severe cases according to the decision of a senior pediatrician. The validated clinical score for acute bronchiolitis were taken after a period of adjustment of at least 5 min and with the child quiet, not crying, without fever, and breathing room air. Respiratory rate were determined by observation of the thoracic movement over a full minute. The degree of accessory muscle use was based on the degree of intercostal or subcostal retraction. Physical examination as well as clinical severity score was recorded for each case at admission and every 12 hours, and at discharge. On discharge, all caregivers of breastfed, partially breastfed and bottle fed infants were advised to continue vitamin D supplementation at dose 400 IU per day

All patients were submitted to careful history taking, complete clinical examination and the following laboratory investigations.

* Complete blood count
* Basal serum vitamin D3 (The 25-hydroxy vitamin D): was done before enrollment of patients in the randomized trial.

Venous blood samples were collected from every subject by sterile venipuncture using disposable syringes. Each sample was then distributed as follows:

1. One ml of blood was disposed into a plastic tube containing EDTA solution for performing complete blood count using electronic cell counter (sysmex kx-21,Japon).
2. |Two ml blood was delivered into plain tube and centrifuged to obtain a clear non hemolyzed serum which was used for performing 25 (OH) vitamin D assays. The specimens were stored at - 20 until the time of the analysis. The serum 25 (OH) D levels were measured using the Enzyme-Linked Immunosorbent Assay (ELISA) method.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 1-24 months of age, diagnosed clinically as acute bronchiolitis and presented with any of the following:

  1. Persistent resting oxygen saturation below 92% in room air.
  2. Marked tachypnea.
  3. Intercostal retractions indicating respiratory distress.
  4. Inability to maintain oral hydration.
  5. Parent unable to care for child at home.

Exclusion Criteria:

1. Infants with history of prematurity (< 37 weeks), chronic cardiopulmonary disease, immunodeficiency, neuromuscular disease, and any other chronic medical condition.
2. Patients receiving any micronutrient supplementation or therapies containing vitamin D for 4 weeks prior to the study period.
3. Infants with previous episodes of wheezing or a physician's diagnosis of asthma.
4. Patients with acute bronchiolitis having very severe clinical score.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | 3 to 5 days
  Length of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: amal osman, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Children's Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842